CLINICAL TRIAL: NCT06290518
Title: Modulation of the Reproductive Microbiota as a Strategy to Increase Rates of Reproductive Success in Couples With Infertility of Unknown Origin
Brief Title: Modulation of Reproductive Microbiota by Ligilactobacillus Salivarius CECT5713
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosearch S.A. (Industry)
Collaborators: Hospital San Carlos, Madrid (Other); Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PROBIFERT P051; NCT05896657 (obsolete NCT alias)
Record Dates: First submitted 2024-02-08; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Infertility Unexplained
Keywords: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Volunteers are classified into 2 groups. All women in the probiotic group consume (oral route) a daily capsule with ~50 mg of freeze-dried probiotic (9.5 log10 CFU of L. salivarius CECT5713; excipient: maltodextrin). All women in the placebo group consume (oral route) a daily capsule with ~50 mg of maltodextrin.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple (Participant, Care Provider, Investigator) Only one person of the collaborator that provides the capsules (Biosearch Life) know the correspondecs between each reference (one reference per each subject) and the arm (probiotic or placebo). The codes are blinded for the participant, the care provider and the investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): All women in the probiotic group consume (oral route) a daily capsule with ~50 mg of freeze-dried probiotic (9.5 log10 CFU of L. salivarius CECT5713; excipient: maltodextrin) during the 6 months prior to the fertility treatment and during the first IVF cycle (estimated 1-2 months). In case of pregnancy, the woman will continue the treatment until 12 weeks of gestation.
  Interventions: Dietary Supplement: Ligilactobacillus salivarius CECT5713
- Placebo group (Placebo Comparator): All women in the placebo group consume (oral route) a daily capsule with ~50 mg of maltodextrin during the 6 months prior to the fertility treatment and during the first IVF cycle (estimated 1-2 months). In case of pregnancy, the woman will continue the treatment until 12 weeks of gestation.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ligilactobacillus salivarius CECT5713 — Oral administration of a capsule containing 9.5 log10 cfu of the strain.
  Arms: Probiotic group
Dietary Supplement: Placebo — Oral administration of a capsule containing maltodextrin.
  Arms: Placebo group

SUMMARY:
The objective of the project is to elucidate if the oral administration of Ligilactobacillus salivarius CECT5713 is capable of improving the rates of term pregnancies in couples with infertility problems of unknown cause. On the other hand, the project is aimed to detect microbiological, immunological and hormonal markers that allow the identification of couples in which the administration of the strain could be particularly effective. This is a randomized, double-blind, parallel-group controlled nutritional intervention study. The intervention (Ligilactobacillus salivarius CECT5713 or placebo) will be performed during the 6 months prior to the fertility treatment and during the first IVF cycle (estimated 1-2 months). In case of pregnancy, the woman will continue the treatment until 12 weeks of gestation.

ELIGIBILITY:
Inclusion Criteria:

* legal age
* Intention to achieve a pregnancy, but without achieving it;
* Be willing to undergo in vitro fertilization treatment;
* Be on the waiting list for the IVF cycle with an expected waiting time > 5 months.

Exclusion Criteria:

* Sterility in one of the members of the couple (azoospermia; impermeability of the fallopian tubes...).
* Genitourinary malformations;
* Concurrence of other severe diseases (e.g.: cancer, AIDS, ALS, morbid obesity...) or uncontrolled diseases (inflammatory bowel diseases, diabetes...).
* Treatment/intervention other than the planned IVF after the start date of the intervention.
* Antibiotic treatment at the start date of the intervention.
* Intention to consume another probiotic supplement in the following 3 months.
* Participation in another clinical trial.
* Allergic/intolerant to the excipient.
* Inability to understand the informed consent form and/or to follow the basic instructions of the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The target is infertility of unknown origin. The outcome is a successful pregnancy.
Enrollment: 72 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Successful pregnancies | 9 months
  Total number of pregnancies with delivery of a healthy baby

SECONDARY OUTCOMES:
Modification of the vaginal microbiota | 9 months
  Variation in the concentration of lactobacilli and other microbes in vaginal samples (Staph ylococcus, Streptococcus, Enterococcus, Corynebacterium, Rothia, Arthrobacter, Acinetobacter, Actinomyces)
Vaginal immunomodulation | 9 months
  Variation in the concentration of immune factors in vaginal samples. The presence and concentration of a wide spectrum of cytokines, chemokines and growth factors (IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12, IL-13, IL-17, G-CSF, GM-CSF, IFN-γ, MCP-1, MIP-1β, RANTES, TGF-β1, 2 and 3, VEGF, GRO-alpha and TNF-alpha)

CONTACTS AND LOCATIONS:
Overall Officials: Juan M. Rodríguez, PhD, Principal Investigator — Complutense University Madrid
Locations (3):
- Spain (3):
  - Biosearch S.A.U., Granada
  - Hospital Clínico San Carlos, Madrid
  - Universidad Complutense de Madrid, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Global and individual reproductive rates, microbiological and immunological data will be available to other researchers once the study (including analyses of all the samples) is completed and published.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: All the raw data will be available to other researchers once the study is published.
Access Criteria: Our intention is that all the raw data will be available as a supplementary tables in an open acess journal. They will be also provided on request.

REFERENCES:
- [Background] Fernandez L, Castro I, Arroyo R, Alba C, Beltran D, Rodriguez JM. Application of Ligilactobacillus salivarius CECT5713 to Achieve Term Pregnancies in Women with Repetitive Abortion or Infertility of Unknown Origin by Microbiological and Immunological Modulation of the Vaginal Ecosystem. Nutrients. 2021 Jan 6;13(1):162. doi: 10.3390/nu13010162. PMID 33419054